CLINICAL TRIAL: NCT01800136
Title: Non-invasive Cortical Stimulation for Pharmacoresistant Neuropathic Pain: rTMS Versus tDCS
Brief Title: Analgesic Effect of Non Invasive Stimulation : Comparison of rTMS and tDCS Efficacy
Acronym: NI-MCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011.662; 2008-A01379-32 (Other: ID-RCB)
Record Dates: First submitted 2012-10-30; First posted 2013-02-27 (Estimated); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Pharmacoresistant Neuropathic Pain
Keywords: pain; neuropathic; cortical stimulation; motor cortex; plasticity; rTMS; tDCS
MeSH Terms: conditions — Pain | interventions — Transcranial Magnetic Stimulation; Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- rTMS; tDCS (Experimental)
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation and Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation and Transcranial Direct Current Stimulation — Five sessions of HF-rTMS or tDCS applied daily during 5 consecutive days

SUMMARY:
The aim of this study is to compare analgesic efficacy of two non invasive techniques based on motor cortex stimulation in neuropathic pain patients. High frequency repetitive transcranial magnetic stimulation (HF-rTMS) of primary motor cortex has been demonstrated to induce an analgesic effect significantly different from placebo; this effect is clinically useful if rTMS sessions are applied daily during five consecutive days. Transcranial direct current stimulation (tDCS) is a new approach of non invasive cortical stimulation but its efficacy in neuropathic pain has been not yet established. The investigators propose to compare the analgesic effect of 5 tDCS sessions applied daily to a similar protocol using HF-rTMS. In parallel to the clinical therapeutic evaluation, functional-MRI will be performed before and after the five sessions of rTMS and tDCS, in order to reveal the potential plasticity induced within motor somatotopic map of the primary motor cortex.

ELIGIBILITY:
Inclusion Criteria:

* patients aged from 18 to 80 years, male or female, fully informed and having given their written consent
* pharmacoresistant neuropathic pain during at least one year, without any change of the pharmacological treatment since at least one month

Exclusion Criteria:

* drug addiction, headache, epilepsy history
* ferromagnetic intracranial device
* implanted stimulator
* absence of contraceptive method for women of childbearing age

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-01-13 (Actual); Primary Completion 2019-06-17 (Actual); Study Completion 2019-06-17 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Pain at the end of the stimulation week Change from Baseline in Pain at the end of the first post-stimulation week Change from Baseline in Pain at the end of the second post-stimulation week | Here the Time Frames : Baseline; 1 week; 2 week; 3 week

SECONDARY OUTCOMES:
objective evaluation of sleep quality | Change from Baseline in percentage of sleep time at the end of the stimulation week; at the end of the first post-stimulation week; and at the end of the of the second post-stimulation week
  actimetry measures
subjective evaluation of sleep quality using a numerical auto-evaluation scale | Change from Baseline in level of tiredness at the end of the stimulation week;at the end of the first post-stimulation week; and at the end of the second post-stimulation week
  the patient is asked to evaluate each day the quality of his sleep using a numerical scale from 0 to 10.
nociceptive and non-nociceptive thresholds | Change from Baseline in nociceptive threshold after the first day of stimulation;after the fifth day of stimulation;Change from Baseline in non-nociceptive threshold after the first day of stimulation;and after the fifth day of stimulation
  Electrical stimulation of variable intensities applied on the hand
evaluation of motor cortex plasticity | Change from Baseline in three-dimensional location of the activation peaks at the end of the stimulation week
  displacement of activation locus found after voluntary movements; comparison of the plastic and analgesic effects of rTMS or tDCS

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Neurologie Fonctionnelle et Epileptologie, Hôpital Neurologique de Lyon et Unité " Intégration Centrale de la Douleur ", 1028 Inserm - UCBL, Lyon, France